CLINICAL TRIAL: NCT00645996
Title: The Influence of Probiotics on the Immunologic Response to Vaccinations in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Ilan Youngster, Assaf Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20070567(101/07)
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Immunity; Measles; Mumps; Rubella
Keywords: Probiotics; vaccines; Measles; Mumps; Rubella
MeSH Terms: conditions — Measles; Mumps; Rubella | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: Probiotics (L.acidophilus and B.lactis)
- 2 (Placebo Comparator): Cornflour
  Interventions: Dietary Supplement: Cornflor

INTERVENTIONS:
Dietary Supplement: Probiotics (L.acidophilus and B.lactis) — 2.1 X 109 L.acidophilus and B.lactis
  Arms: 1
Dietary Supplement: Cornflor — Cornflour 2 gram daily
  Arms: 2

SUMMARY:
Background: It is well established that the presence of bacteria in the intestine has a profound influence on health. Probiotics, ("beneficial bacteria") have shown ameliorating effects on various infectious diseases. The influence of probiotics on several immune-mediated conditions has also been investigated, among them, atopic dermatitis ("Asthma of the skin"), and milk allergy.

The precise mechanism of action of probiotics is not fully understood. Several animal and human studies have shown the probiotic bacteria to influence the immune system. The aim of the present study is to evaluate whether supplementing the diet with oral probiotics affects the immune response of children following routine vaccination against 4 common childhood viral diseases: Mumps, Measles, Rubella and Varicella.

Objective(s) and Hypothesis(es):

Hypothesis: Administration of probiotics will increase the amount of antibodies produced following vaccination for Measles, Mumps, Rubella and Varicella, by over 15%.

Objectives:

* To determine whether administration of probiotics during infancy influences antibody levels following the routine childhood vaccinations.
* To determine whether administration of probiotics during infancy influences the rate of adverse effects following the routine childhood vaccinations.

Potential Impact: Vaccines, alongside with the discovery of Penicillin, have been cited as the great public health successes of the 20th century. However, even in countries with maximal childhood immunization coverage, the protective effect is not optimal. For example, only 70% to 90% of children immunized against chickenpox are actually protected against the disease. If we succeed in raising these numbers, even by a single percent, it will have a huge impact on society.

ELIGIBILITY:
Inclusion Criteria:

* Age: 9-11 months.
* Parent or guardian intending to follow the recommended immunization schedule in Israel.
* Parent or guardian possessing sufficient knowledge of the Hebrew language.

Exclusion Criteria:

* Infants suffering from any chronic diseases / conditions resulting in immune depression.
* Infants taking medications affecting the immune system.
* Infants with permanent invasive catheters.
* Infants born prematurely (prior to gestational week 35)
* Parent or guardian objecting to collection of blood sample at the end of study.

Ages: 9 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-07 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
The level of antibodies against Measles, Mumps, Rubella and Varicella in the study group compared to the placebo group. | 1 year

SECONDARY OUTCOMES:
The number of vaccine-related adverse events in the study group compared to the placebo group. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eran Kozer, Principal Investigator — Assaf Harofeh MC; Ilan Youngster, MD, Principal Investigator — Assaf Harofeh MC
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel